CLINICAL TRIAL: NCT01226550
Title: Treatment of Primary Peritoneal Carcinosis of Digestive Origin Using Cytoreductive Surgery and Hyperthermic Intraoperative Peritoneal Chemotherapy With Mitomycin C and Irinotecan
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004.368
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Peritoneal Carcinosis (PC)
Keywords: hyperthermic intraoperative peritoneal chemotherapy (HIPEC); Irinotecan; Pharmacokinetics; peritoneal carcinomatosis (PC)
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Cytoreduction Surgical Procedures; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cytoreductive surgery and HIPEC (Experimental)
  Interventions: Procedure: cytoreductive surgery and HIPEC

INTERVENTIONS:
Procedure: cytoreductive surgery and HIPEC — The most complete cytoreductive surgery possible (ideally macroscopically complete) followed by a closed-abdomen hyperthermic intraoperative peritoneal chemotherapy (HIPEC), using a closed circuit connected to the self-regulating Cavitherm machine (EEC certified). This perfusion apparatus records temperature, flow, and pressure for 90 minutes at real temperature (42-43°C).
  The dialysate is made up of peritoneal dialysis fluid containing 0.7 mg/kg of MMC and increasing doses of irinotecan added to the dialysate the last 30 minutes of the HIPEC.
  Potentiation of irinotecan using an intravenous FUFOL perfusion at least 1hour before HIPEC (1st dose level: 10 mg/m² of folinic acid, then 200 mg/m² of 5-FU; 2nd dose level: 20 mg/m² of folinic acid, then 400 mg/m² of 5-FU).

SUMMARY:
This is an open, non-randomized, phase I-II, pilot study, which evaluates the combination of optimum cytoreductive surgery and hyperthermic intraoperative peritoneal chemotherapy (HIPEC) with mitomycin C (MMC) and irinotecan. The latter drug will be administered in escalating doses to patients with gastric, colorectal, appendicular, or primary peritoneal carcinosis (PC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a peritoneal carcinosis (PC) either of digestive origin or primary: a colorectal or gastric carcinosis, a peritoneal pseudomyxoma or mesothelioma, or a primary carcinosis of the peritoneum regardless the number of prior treatment lines.
* A PC and primary tumor considered to be resectable according to preoperative clinical and paraclinical data: absence of mesenteric retraction and absence of bladder invasion.
* Patients in good general health (ASA ≤ 2).
* Absence of cardiorespiratory failure (PaO2 > 60 mmHg in a stable condition, dyspnea ≤ NYHA stage 1, left ventricular ejection fraction > 60%.).
* Prothrombin level >70 %, total bilirubin < 2 x the normal level, ASAT and ALAT < 2.5 x normal levels, and alkaline phosphatases < 5 x normal levels.
* Creatinine clearance > 60 ml/min, polynuclear neutrophils > 1500/mm3, and a white blood cell count > 4000 /mm3.
* Patients who give written, informed consent.
* Patients affiliated with the French universal healthcare system.

Exclusion Criteria:

* Patients with a PC with ovarian, mammary, biliary, pancreatic, or bronchial origin.
* Evolutive patients after systemic chemotherapy.
* Patients with a PC considered to be irresectable according to preoperative clinical and paraclinical data: mesenteric retraction or bladder invasion.
* Patients in poor general health (ASA > 2).
* Cardiorespiratory failure (dyspnea > NYHA stage 1, PaO2 < 60 mmHg in a stable condition)
* Prothrombin level < 70 %.
* Any brain abnormality showing on the head scan.
* Signs of heart failure and especially left ventricular ejection fraction < 60% on the cardiac ultrasound.
* Thrombocytopenia < 100 000 / mm3
* Visceral metastases other than a single resectable liver metastasis.
* Pregnancy or breast feeding.
* Chronic inflammatory intestinal disease and/or an intestinal obstruction.
* History of severe hypersensitivity to irinotecan hydrochloride trihydrate or one of the excipients of Campto.
* Bilirubinemia > 3 times the normal upper limit
* Yellow fever vaccine.
* Prophylactic treatment with phenytoin.
* Severe medullary insufficiency.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Morbidity rate | 30 days postoperative
  postoperative complications (class III and IV, Common Terminology Criteria V3; National Cancer Institute)

SECONDARY OUTCOMES:
Mortality rate | 30 days postoperative
Intraperitoneal and serumal concentration (pharmacokinetics) of mitomycine C, irinotecan, and its metabolites. | per-HIPEC
  Plasma, peritoneal, and urinary values for MMC, irinotecan, SN-38, SN-38G, APC, and NPC.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Générale et Thoracique, Centre Hospitalier Lyon-Sud, Pierre-Bénite, France

REFERENCES:
- [Result] Cotte E, Passot G, Tod M, Bakrin N, Gilly FN, Steghens A, Mohamed F, Glehen O. Closed abdomen hyperthermic intraperitoneal chemotherapy with irinotecan and mitomycin C: a phase I study. Ann Surg Oncol. 2011 Sep;18(9):2599-603. doi: 10.1245/s10434-011-1651-1. Epub 2011 Mar 19. PMID 21424369